CLINICAL TRIAL: NCT04366427
Title: Effects of Enriched Oxygen Mixtures and Exercise on Oxidative Stress and Stem Cells Proliferation in Athletes.
Brief Title: Enriched Oxygen Mixtures in Athletes
Acronym: OXY-SPORT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: Performa di Crocicchia Srl (Unknown)
Responsible Party: Principal Investigator, Gerardo Bosco, Associate Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HEC-DSB/04-19
Record Dates: First submitted 2020-03-04; First posted 2020-04-28 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Oxidative Stress; Stem Cell Research
Keywords: Hyperbaric Oxigenation; Sport Medicine; Training; Recovery; Oxidative Stress; Stem Cell Research

STUDY DESIGN:
Intervention Model Description: Five arms: one control without treatment; one at low pressure (1.45 ATA); one at standard pressure (2.5 ATA); one at atmospheric pressure (1 ATA) breathing air mixture with 30% O2; one at atmospheric pressure (1 ATA) breathing air mixture with 50% O2;
Who Masked: Outcomes Assessor
Masking Description: Participants, Care Provider, and Investigators will not be masked. Only outcome assessors will only evaluate data without knowing the arm the patients were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Low-pressure hyperbaric oxygenation (L-HBO) (Experimental): Low-pressure hyperbaric oxygen administration at 1.45 ATA for 60 minutes, inclusive of compression and decompression times, and a 3-minute air pause at the midtime. For a total of 20 sessions (3-4 per week).
  Interventions: Combination Product: L-HBO
- Standard-pressure hyperbaric oxygenation (HBO) (Experimental): Standard pressure hyperbaric oxygen administration at 2.5 ATA for 60 minutes, inclusive of compression and decompression times, and a 3-minute air pause at the midtime. For a total of 20 non-consecutive sessions (3-4 per week).
  Interventions: Combination Product: HBO
- Control (No Intervention): Control group of athletes, no intervention.
- 30% O2 (Experimental): Administration of air mixture with 30% O2, subjects breathing this mixture for 60 minutes for a total of 20 non-consecutive sessions (3-4 per week).
  Interventions: Combination Product: 30% O2
- 50% O2 (Experimental): Administration of air mixture with 50% O2, subjects breathing this mixture for 60 minutes for a total of 20 non-consecutive sessions (3-4 per week).
  Interventions: Combination Product: 50% O2

INTERVENTIONS:
Combination Product: L-HBO — as previously described.
  Other Names: Low Pressure Oxygenation
  Arms: Low-pressure hyperbaric oxygenation (L-HBO)
Combination Product: HBO — as previously described.
  Other Names: Standard Pressure Oxygenation
  Arms: Standard-pressure hyperbaric oxygenation (HBO)
Combination Product: 30% O2 — as previously described
  Other Names: 30% O2 mixture
  Arms: 30% O2
Combination Product: 50% O2 — as previously described
  Other Names: 50% O2 mixture
  Arms: 50% O2

SUMMARY:
Currently, Hyperbaric Oxigen (HBO) is a widely used treatment for several conditions. There are 14 indications for HBO, officially recognized by the Undersea and Hyperbaric Medical Society (UHMS), but research is discovering other interesting applications.

HBO plays an important role in enhancing antioxidant defense mechanisms by increasing radical oxygen species (ROS) and nitric oxide species (NOS). This controlled oxidative stress has been shown to stop the vicious circle of inflammation - damage - hypoxia already seen in several diseases. Increased neoangiogenesis has been demonstrated at pressures of 2 atmospheres absolute (ATA), while effects helping ischemic tissues need pressures between 2.5 and 2.8 ATA to develop. Also, stem cell proliferation and mobilization have been demonstrated after HBO treatments.

During sports activities, metabolism generates waste products - mostly CO2, lactic acid, but also ROS. HBO could be useful in modulating antioxidant mechanisms and increasing stem cell mobilization, thus helping cells in the recovery after training and sportive competitions.

The authors hypothesize that:

1. HBO can reduce oxidative stress and induce stem cell mobilization in healthy professional athletes;
2. hyperoxic mixtures can reduce oxidative stress and induce stem cells mobilization in healthy professional athletes;
3. HBO at low pressures (L-HBO at 1.45 ATA) is at least comparable to conventional HBO (at 2.5 ATA) in reducing oxidative stress and increasing stem cell mobilization.

The Authors will include healthy athletes. These will be randomly assigned to a control group, a L-HBO group, a HBO group, a 30% O2 group, or a 50% O2 group.

The Authors will assess oxidative stress changes and stem cells proliferation before and after 20 L-HBO/HBO/30% O2 mix/50% O2 mix treatments, and after 2 months after the end of treatments.

DETAILED DESCRIPTION:
Subjects will be recruited through public announcements in local gyms and gathered to explain the protocol. Those willing to participate will sign a written informed consent and recruited. To be included, all the subjects will undergo a general medical screening to allow hyperbaric treatments. This will include weight, height, non-invasive arterial blood pressure, and heart rate measurements.

After inclusion, subjects will be randomly assigned to three arms using an electronic number generator by personnel not directly involved in the experiment:

* Arm 1(control): no intervention.
* Arm 2 (L-HBO): treated with oxygen at 1.45 ATA for 60 min (inclusive of compression and decompression times, and an air break of 3 minutes breathing air);
* Arm 3 (HBO): treated with oxygen at 2.5 ATA for 60 min (inclusive of compression and decompression times, and an air break of 3 minutes breathing air).
* Arm 4 (30% O2): breathing an air mixture with 30% of oxygen at atmospheric pressure (1 ATA).
* Arm 5 (50% O2): breathing an air mixture with 50% of oxygen at atmospheric pressure (1 ATA).

Subjects included in Arm 2, 3, 4, 5 will undergo a total of 20 treatments. They will follow a personalized diet proportional to their energetic expenditure.

The Authors will identify 3 time-points in the protocol:

TIME 0 (T0): immediately after inclusion, before any treatment or experiment; TIME 1 (T1): at the end of HBO treatments; TIME 2 (T2): 2 months after the end of HBO treatments.

The following exams will be performed on the included subjects:

* a standardized panel including Complete Blood Count (CBC), creatinine, Blood Urea Nitrogen (BUN), C reactive protein, and VES will be performed at T0, T1, and T2.
* oxidative stress markers will be analyzed on blood, urine, and saliva samples. On blood samples (T0; T1; T2), the Authors will measure IL-1 beta, IL-6, TNF-alfa, reactive oxygen species and total antioxidant capacity (by paramagnetic resonance), total (tot) and reduced (red) aminothiols (by fluorescence spectroscopy), 3-nitrotyrosine (3-NT) (by competitive immunoassay).

On urine samples (T0; T1; T2), the Authors will assess lipid peroxidation by measuring 8-isoprostane concentration (by competitive immunoassay), nitrite and nitrate (NO2/NO3) concentration (by colorimetry based on the Griess reaction), inducible Nitric Oxide Synthase (by ELISA commercially available kit), creatinine, neopterine, and uric acid concentrations, 8-oh-2-deoxyguanosine (by competitive immunoassay).

On saliva samples (T0; T1; T2) the Authors will measure reactive oxygen species and total antioxidant capacity (by paramagnetic resonance), and cortisol (by competitive immunoassay).

* stem cells will be analyzed on blood samples (at T0, T1, T2) (by flow cytometry).

Blood samples (approximately 6-12 ml) will be drawn from the veins of the forearms (preferentially on the non-dominant limb); plasma and erythrocytes will be separated by centrifuge at 1000×g for 10 min at 4°C. Urine samples will be collected by voluntary voiding in sterile containers. 1 mL of saliva will be obtained by Salivette devices (Sarstedt, Nümbrecht, Germany). The subjects will be instructed to refrain from drinking, eating, smoking, brushing their teeth, and using mouthwash in the 30 min before salivary collection.

All samples will be stored in multiple aliquots at - 80 °C until assayed and thawed only once before analysis.

With this setting, blinding of patients and investigators will be impossible due to different structural characteristics. However, outcome assessors will be blinded to patients' allocation.

ELIGIBILITY:
Inclusion Criteria:

* professional athletes
* performing at least 3 training sessions/week

Exclusion Criteria:

* previous pneumothorax
* problems with compensation maneuvers
* known epilepsy
* active smoker

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Reactive oxygen species production | On blood and saliva: at baseline (T0), at the completion of treatments (Time 1: 5 weeks after the baseline) and 2 months after the end of treatments (Time 2)
  Reactive oxygen species production (μmol min-1) (by paramagnetic resonance)
Change in Total antioxidant capacity | On blood and saliva: at baseline (T0), at the completion of treatments (Time 1: 5 weeks after the baseline) and 2 months after the end of treatments (Time 2)
  Total antioxidant capacity (by paramagnetic resonance) (mM)
Change in Cortisol levels | On saliva: at baseline (T0), at the completion of treatments (Time 1: 5 weeks after the baseline) and 2 months after the end of treatments (Time 2)
  Cortisol (by competitive immunoassay) (ng/ml)
Change in nitrite and nitrate (NO2/NO3) concentration | On urine: at baseline (T0), at the completion of treatments (Time 1: 5 weeks after the baseline) and 2 months after the end of treatments (Time 2)
  nitrite and nitrate (NO2/NO3) concentration (by colorimetry based on the Griess reaction) (μM)
Change in inducible Nitric Oxide Synthase (iNOS) | On urine: at baseline (T0), at the completion of treatments (Time 1: 5 weeks after the baseline) and 2 months after the end of treatments (Time 2)
  inducible Nitric Oxide Synthase (by ELISA commercially available kit) (IU mL-1)
Change in aminothiols levels | On blood: Change from Baseline (T0) aminothiols concentration after the exercise test (Time 1: the day after baseline measurements), and at the completion of treatments after a second exercise test (Time 3: 5 weeks after the baseline)
  total (tot) and reduced (red) aminothiols (by fluorescence spectroscopy) (μmol L-1)
Change in Cytokines levels | On blood: at baseline (T0), at the completion of treatments (Time 1: 5 weeks after the baseline) and 2 months after the end of treatments (Time 2)
  IL-1 beta, IL-6, TNF-alfa (pg ml-1)
Change in lipid peroxidation markers | On urine: at baseline (T0), at the completion of treatments (Time 1: 5 weeks after the baseline) and 2 months after the end of treatments (Time 2)
  On urine samples, we will assess lipid peroxidation by measuring 8-isoprostane and 8-OH-deoxyguanosine concentration (by competitive immunoassay) - (pg mg-1 creatinine)
Change in Renal damage markers | On urine: at baseline (T0), at the completion of treatments (Time 1: 5 weeks after the baseline) and 2 months after the end of treatments (Time 2)
  On urine samples, we will assess renal damage by measuring creatinine (g-L-1), neopterin (μmol·mol-1 creatinine), and uric acid levels (mg/dl).
Change in 3-nitrotyrosine levels | On urine: at baseline (T0), at the completion of treatments (Time 1: 5 weeks after the baseline) and 2 months after the end of treatments (Time 2)
  3-nitrotyrosine (3-NT) (by competitive immunoassay)( nM·L-1)
Change in Stem cells mobilization | On blood: at baseline (T0), at the completion of treatments (Time 1: 5 weeks after the baseline) and 2 months after the end of treatments (Time 2)
  Stem cells (by flow cytometry) (%)

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Bosco, MD, PhD, Principal Investigator — University of Padova; Matteo Paganini, MD, Study Director — University of Padova
Locations (1):
- Human Physiology Institute, Department of Biomedical Sciences, University of Padova, Padua, Veneto, Italy

IPD SHARING:
Plan to Share IPD: No
First, data will be shared with the funding partner and disseminated through publications and meetings, and then made available upon request.

REFERENCES:
- [Background] Pedoto A, Nandi J, Yang ZJ, Wang J, Bosco G, Oler A, Hakim TS, Camporesi EM. Beneficial effect of hyperbaric oxygen pretreatment on lipopolysaccharide-induced shock in rats. Clin Exp Pharmacol Physiol. 2003 Jul;30(7):482-8. doi: 10.1046/j.1440-1681.2003.03865.x. PMID 12823263
- [Background] Bosco G, Yang ZJ, Nandi J, Wang J, Chen C, Camporesi EM. Effects of hyperbaric oxygen on glucose, lactate, glycerol and anti-oxidant enzymes in the skeletal muscle of rats during ischaemia and reperfusion. Clin Exp Pharmacol Physiol. 2007 Jan-Feb;34(1-2):70-6. doi: 10.1111/j.1440-1681.2007.04548.x. PMID 17201738
- [Background] Yang ZJ, Xie Y, Bosco GM, Chen C, Camporesi EM. Hyperbaric oxygenation alleviates MCAO-induced brain injury and reduces hydroxyl radical formation and glutamate release. Eur J Appl Physiol. 2010 Feb;108(3):513-22. doi: 10.1007/s00421-009-1229-9. Epub 2009 Oct 23. PMID 19851780
- [Background] Bosco G, Yang ZJ, Di Tano G, Camporesi EM, Faralli F, Savini F, Landolfi A, Doria C, Fano G. Effect of in-water oxygen prebreathing at different depths on decompression-induced bubble formation and platelet activation. J Appl Physiol (1985). 2010 May;108(5):1077-83. doi: 10.1152/japplphysiol.01058.2009. Epub 2010 Feb 25. PMID 20185629
- [Background] Morabito C, Bosco G, Pilla R, Corona C, Mancinelli R, Yang Z, Camporesi EM, Fano G, Mariggio MA. Effect of pre-breathing oxygen at different depth on oxidative status and calcium concentration in lymphocytes of scuba divers. Acta Physiol (Oxf). 2011 May;202(1):69-78. doi: 10.1111/j.1748-1716.2010.02247.x. Epub 2011 Mar 1. PMID 21199400
- [Background] Nasole E, Nicoletti C, Yang ZJ, Girelli A, Rubini A, Giuffreda F, Di Tano A, Camporesi E, Bosco G. Effects of alpha lipoic acid and its R+ enantiomer supplemented to hyperbaric oxygen therapy on interleukin-6, TNF-alpha and EGF production in chronic leg wound healing. J Enzyme Inhib Med Chem. 2014 Apr;29(2):297-302. doi: 10.3109/14756366.2012.759951. Epub 2013 Jan 30. PMID 23360079
- [Background] Camporesi EM, Bosco G. Mechanisms of action of hyperbaric oxygen therapy. Undersea Hyperb Med. 2014 May-Jun;41(3):247-52. PMID 24984320
- [Background] Bosco G, Vezzani G, Mrakic Sposta S, Rizzato A, Enten G, Abou-Samra A, Malacrida S, Quartesan S, Vezzoli A, Camporesi E. Hyperbaric oxygen therapy ameliorates osteonecrosis in patients by modulating inflammation and oxidative stress. J Enzyme Inhib Med Chem. 2018 Dec;33(1):1501-1505. doi: 10.1080/14756366.2018.1485149. PMID 30274530
- [Background] Moskowitz A, Andersen LW, Huang DT, Berg KM, Grossestreuer AV, Marik PE, Sherwin RL, Hou PC, Becker LB, Cocchi MN, Doshi P, Gong J, Sen A, Donnino MW. Ascorbic acid, corticosteroids, and thiamine in sepsis: a review of the biologic rationale and the present state of clinical evaluation. Crit Care. 2018 Oct 29;22(1):283. doi: 10.1186/s13054-018-2217-4. PMID 30373647
- [Background] Fisher-Wellman K, Bloomer RJ. Acute exercise and oxidative stress: a 30 year history. Dyn Med. 2009 Jan 13;8:1. doi: 10.1186/1476-5918-8-1. PMID 19144121
- [Background] Menzies P, Menzies C, McIntyre L, Paterson P, Wilson J, Kemi OJ. Blood lactate clearance during active recovery after an intense running bout depends on the intensity of the active recovery. J Sports Sci. 2010 Jul;28(9):975-82. doi: 10.1080/02640414.2010.481721. PMID 20544484
- [Background] Van Hooren B, Peake JM. Do We Need a Cool-Down After Exercise? A Narrative Review of the Psychophysiological Effects and the Effects on Performance, Injuries and the Long-Term Adaptive Response. Sports Med. 2018 Jul;48(7):1575-1595. doi: 10.1007/s40279-018-0916-2. PMID 29663142